CLINICAL TRIAL: NCT04234698
Title: Patient Characteristics, Treatment Patterns and Incidence of Events (Discontinuation, Persistence, Key Primary Clinical Outcomes) in NVAF Patients Initiating OAC Therapy in Colombia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661148
Record Dates: First submitted 2019-12-20; First posted 2020-01-21 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
Keywords: oral anticoagulants; apixaban; rivaroxaban; dabigatran; warfarin; non valvular atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aim to assess demographic and clinical characteristics , treatment patterns and as exploratory analysis will descriptively assess the time to clinical events of NVAF patients treated with oral anticoagulants (OACs) in Colombia through observational, descriptive study of a retrospective cohort of adult patients diagnosed with NVAF in selected Health Maintenance Organizations (HMO) of Colombia. The information will be used in the study comes exclusively form secondary sources: claim databases and medical records.

DETAILED DESCRIPTION:
The study has the following primary objectives:

* To assess demographic and clinical characteristics of NVAF patients treated with oral anticoagulants (OACs) in Colombia.
* To describe treatment patterns (eg OAC usage,dose, concomitant medications, persistance)

And as exploratory analysis to descriptively assess the time to clinical events (Effectiveness and Safety Outcomes) among patients persistent on OAC therapy

It is an observational, descriptive study of a retrospective cohort of adult patients diagnosed with NVAF in selected Health Maintenance Organizations (HMO) of Colombia. These patients will be identified from the drug claim database, whose index date of the study will be the first prescription with any of the oral anticoagulants, that is, they are patients with NVAF for the first time starting a therapy with any of the NOACs between January 1, 2013 and June 30, 2018 and follow up period will be among January 2013 to July 2019, to ensure that the last patients can provide follow-up for one year. Patients will be required to have an NVAF diagnosis before or on the index date and health plan for 6 months pre-index date (baseline period). Colombia. The information will be used in the study comes exclusively form secondary sources: claim databases and medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AF considered according to the following diagnoses as per the 10th revision of the International classification of diseases (ICD-10) I48 codes at some point before or on the index date, without recorded valvular disease;
* Patients who have started treatment with apixaban, dabigatran, rivaroxaban and warfarin for the first time during the identification period, understanding as start of drug delivery by insurer, and after the diagnosis of AF between January 1, 2013 to June 30, 2018;
* Patients starting apixaban, dabigatran, rivaroxaban from January 1, 2013 to June 30, 2018 in patients previously exposed to warfarin;
* Patient had continuous health plan enrolment for 6 months pre-index date (baseline period);
* Patients older than 18 years old on the index date;
* NVAF diagnosis before or on the index date.

Exclusion Criteria:

* Patients with any of the following diagnoses prior to the use of the treatments of interest or index date:

  * Valvular heart disease or valve replacement - ICD-10 codes: I05, I06, I07, I08, I09, I21, I22, I34, I35, I36, I37, I38, I39, I700, I702-I709; Q22, Q23, Q25, T82, Z95
  * Pregnancy during the study period. ICD-10 O00-O9A
  * Diagnosis of venous thromboembolism (VTE) - ICD-10 codes: I26, I80 - I82;
* Individuals with a transitory diagnosis of NVAF prior to the use of the treatments of interest or index date;
* Exposure to more than one OAC on or after the index date, during the follow-up period;
* NOAC doses different from those recommended by the manufacturing laboratories.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total population of patients treated with any oral anticoagulant between January 1, 2013 and June 30, 2018 will be analyzed in the claim database. This means that patients who start warfarin and NOACs would be included within this period. Patients who initiate NOACs within the established period and who have been exposed to warfarin before 2013 will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 2076 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with non-valvular atrial fibrillation (NVAF) who initiated treatment with warfarin and any of new oral anticoagulants (NOACs) [dabigatran, rivaroxaban, apixaban] between 01-January-2013 to 30-June-2018,registered in Health Maintenance Organizations(HMO)of Colombia were observed retrospectively. Data was retrieved from claim database and medical records during approximately 2 months of this study.
Pre-assignment Details: Baseline for this study was 6 months prior to the index date. The index date was the date of first prescription with any of the oral anticoagulants (OACs).
Groups:
- Warfarin: Participants diagnosed with NVAF who initiated treatment with warfarin between 01-January-2013 to 30-June-2018 were observed in this retrospective study. Participants were followed up until July 2019.
- NOACs: Participants diagnosed with NVAF, who initiated treatment with any of the NOACs (dabigatran, rivaroxaban and apixaban) between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated NOACs between 01-January-2013 and 30-June-2018 were also included. Participants were followed up until July 2019.
Period: Overall Study
Arm/Group | Warfarin | NOACs
Started | 459 | 1617
Completed | 459 | 1617
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants diagnosed with NVAF who initiated treatment with warfarin and NOACs between 01-January-2013 to 30-June-2018 or who were exposed to warfarin before 2013 and initiated treatment with NOACs within the established period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin | NOACs | Total
Number analyzed (Participants) | 459 | 1617 | 2076
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.6 (10.0) | 73.7 (10.0) | 73.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258 | 926 | 1184
  Male | 201 | 691 | 892
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and Ethnicity were not collected from any participant. Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: Centimeters] | 160.4 (10.2) | 160.9 (9.9) | 160.8 (10.0)
Weight [Mean (Standard Deviation); unit: Kilograms] | 70.0 (14.0) | 70.7 (14.4) | 70.0 (14.0)
Number of Participants According to Geographic Regions [Count of Participants; unit: Participants]
  Bogota/center | 175 | 497 | 672
  Atlantic Coast | 35 | 486 | 521
  Coffee belt | 122 | 202 | 324
  Santander | 48 | 146 | 194
  Antioquia | 60 | 128 | 188
  Center-West | 16 | 133 | 149
  Eastern plains | 3 | 25 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms per meter square] | 27.1 (4.9) | 27.3 (5.0) | 27.3 (4.9)
Number of Participants With Alcohol Intake at OAC Prescription Date [Count of Participants; unit: Participants] | 5 | 10 | 15
Number of Participants With History of Comorbidities at Index Date [Count of Participants; unit: Participants]
  Ischemic or Hemorrhagic Stroke | 56 | 263 | 319
  Gastrointestinal Bleeding | 5 | 20 | 25
  Intracranial Bleeding | 0 | 6 | 6
  Transient Ischemic Attack | 4 | 27 | 31
  Thromboembolism | 0 | 0 | 0
  Other bleeding | 1 | 12 | 13
Number of Participants With Bleeding History or Predisposition to Bleeding at Start of OAC Treatment [Count of Participants; unit: Participants] | 1 | 12 | 13
Number of Participants With International Normalized Ratio(INR)Greater Than(>)60%: Start OAC Therapy [Count of Participants; unit: Participants] — Population: INR was evaluated only for participants who were exposed to warfarin.
  Participants
    number analyzed (Participants) | 459 | 0 | 459
    (all) | 134 | 0 | 134

OUTCOME MEASURES:

1. Primary Outcome: Time to Diagnose NVAF by Each OAC Treatment
Description: Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Days
Groups:
- NOACs - Rivaroxaban: Participants diagnosed with NVAF, who initiated treatment with rivaroxaban between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated rivaroxaban between 01-January-2013 and 30-June-2018 were also included. Participants were followed up until July 2019.
- NOACs - Apixaban: Participants diagnosed with NVAF, who initiated treatment with apixaban between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated apixaban between 01-January-2013 and 30-June-2018 were also included. Participants were followed up until July 2019.
- NOACs - Dabigatran: Participants diagnosed with NVAF, who initiated treatment with dabigatran between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated dabigatran between 01-January-2013 and 30-June-2018 were also included. Participants were followed up until July 2019.
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 459 | 950 | 405 | 262
Days | 71 (230.8) | 324 (712.2) | 218 (541.2) | 406 (676.0)

2. Primary Outcome: Number of Participants With Comorbidities
Description: Participants classified according to the comorbidities they had were reported in this outcome measure. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018. One participant may have more than one comorbidity.
Time Frame: From index date until switch of treatment, discontinuation, death, first stroke/systemic embolism, or major bleeding, or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants
  Diabetes Mellitus | 100 | 370
  Liver Disease | 5 | 25
  Hypertension | 386 | 1430
  Rheumatic disease | 23 | 58
  Acquired Immune Deficiency Syndrome (AIDS) | 0 | 0
  Chronic Kidney Disease | 196 | 892
  Moderate Renal Disease | 163 | 661
  Congestive Heart Failure | 86 | 231
  Acute Myocardial Infarction | 70 | 308
  Chronic Obstructive Pulmonary Disease (COPD) | 84 | 276
  Peripheral Vascular Disease | 30 | 73
  Dementia | 11 | 48
  Hemiplegia | 9 | 38
  Connective Tissue Disease | 23 | 58
  Leukemia and Lymphoma | 2 | 9
  Peptic Ulcer Disease | 4 | 7
  Metastatic Solid Tumor (Cancer) | 0 | 21
  Acute myocardial infarction | 70 | 308

3. Primary Outcome: Number of Participants With Uncontrolled Hypertension at OAC Prescription Date
Description: as for outcome 1
Time Frame: At index date (any time between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 19 | 50

4. Primary Outcome: Number of Participants With Use of Aspirin at Start OAC Treatment
Description: as for outcome 1
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 191 | 660

5. Primary Outcome: Number of Participants With Use of Clopidogrel at Start of OAC Treatment
Description: as for outcome 1
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 37 | 133

6. Primary Outcome: Number of Participants With Use of Non-Steroidal Anti-Inflammatory Drugs at Start of OAC Treatment
Description: Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018. In this study Aspirin was not considered as NSAID due to doses used in Colombia.
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 18 | 50

7. Primary Outcome: HAS-BLED Score at Start of OAC Treatment
Description: The risk of bleeding in participants was assessed using Hypertension, Abnormal renal and liver function, Stroke, Bleeding, Labile INR, Elderly, (age >65 years), Drugs or alcohol (HAS-BLED) score. Score ranged from 0 to 8 with higher scores indicating greater risk of bleeding. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Units on a scale | 2.25 (0.95) | 1.99 (0.90)

8. Primary Outcome: CHA2DS2-VASc Score at Start of OAC Treatment
Description: The CHA2DS2-VASc scale is an evaluation of stroke risk in participants with atrial fibrillation. CHA2DS2-VASc is the Congestive heart failure, Hypertension, Age (> 75), Diabetes mellitus, Stroke/TIA, Vascular disease, Age 65-74, Sex Category score , with total scores ranging from 0 to 9, with low scores indicating low risk for stroke, and high scores indicating high risk for stroke. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Units on a scale | 3.6 (1.5) | 3.6 (1.5)

9. Primary Outcome: Number of Participants With Anemia at Start of OAC Treatment
Description: as for outcome 1
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 62 | 217

10. Primary Outcome: Number of Participants With Stroke
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 56 | 263

11. Primary Outcome: Duration of Follow-up in Participants With Stroke
Description: as for outcome 1
Time Frame: as for outcome 2
Population: Analysis population included all eligible participants diagnosed with NVAF who initiated treatment with warfarin and NOACs between 01-January-2013 to 30-June-2018 or who were exposed to warfarin before 2013 and initiated treatment with NOACs within the established period. Here ''Overall Number of Participants Analyzed'' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 56 | 263
Days | 244 (157) | 680 (559)

12. Primary Outcome: Number of Participants According to Type of Stroke
Description: Number of participants with type of stroke classified as either ischemic cerebrovascular event or hemorrhagic cerebrovascular event were reported in this outcome measure. Participants who reported cerebral infarction, stroke: not specified as hemorrhage or infarction in their medical history during the follow-up period were classified under ischemic cerebrovascular event and participants who reported subarachnoid hemorrhage, intracerebral hemorrhage and other nontraumatic intracranial hemorrhage in their medical record were classified under hemorrhagic stroke. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 56 | 263
Participants
  Ischemic cerebrovascular event | 11 | 45
  Hemorrhagic cerebrovascular event | 5 | 2

13. Primary Outcome: Number of Participants With Pulmonary Embolism
Description: The number of participants who had pulmonary embolism were reported in this outcome measure. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 1 | 5

14. Primary Outcome: Duration of Follow-up in Participants With Pulmonary Embolism
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 1 | 5
Days | 25 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 620 (409)

15. Primary Outcome: Number of Participants With Gastrointestinal Bleeding
Description: The number of participants who had gastrointestinal bleeding were reported in this outcome measure. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 19 | 23

16. Primary Outcome: Duration of Follow-up in Participants With Gastrointestinal Bleeding
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 19 | 23
Days | 501 (561) | 444 (298)

17. Primary Outcome: Number of Participants With Intracranial Bleeding
Description: The number of participants who had intracranial bleeding were reported in this outcome measure. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 5 | 2

18. Primary Outcome: Duration of Follow-up in Participants With Intracranial Bleeding
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 5 | 2
Days | 400 (355) | 206 (228)

19. Primary Outcome: Number of Deaths
Description: as for outcome 1
Time Frame: From index date until death or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 1 | 5

20. Primary Outcome: Duration of Follow-up in Participants Who Died
Description: as for outcome 1
Time Frame: as for outcome 19
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 1 | 5
Days | 881 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed. | 722 (742)

21. Primary Outcome: Time Under OAC Treatment (Persistence) by Each OAC Treatment
Description: Persistence was defined as the time under each OAC treatment, calculated as the time in days from the index date to the date of discontinuation or change of treatment. Participants were censored at the end of their follow-up period. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: From index date until switch of treatment, discontinuation, or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 459 | 950 | 405 | 262
Days | 440 [158 to 805] | 491 [181 to 985] | 364 [202 to 627] | 608 [279 to 1176]

22. Primary Outcome: Number of Participants With Other Major Bleeding
Description: The number of participants who had other major bleeding were reported in this outcome measure. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 17 | 19

23. Primary Outcome: Duration of Follow-up in Participants With Other Major Bleeding
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 17 | 19
Days | 233 (385) | 585 (631)

24. Primary Outcome: Dose of Initial OAC Prescription by Each OAC Treatment
Description: as for outcome 1
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 459 | 950 | 405 | 262
Milligrams | 4.5 (2.6) | 17.9 (2.7) | 7.8 (2.5) | 239 (48.5)

25. Primary Outcome: Number of Doses Dispensed at Initial OAC Treatment by Each OAC Treatment
Description: as for outcome 1
Time Frame: At index date (anytime between 01-January-2013 to 30-June-2018)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Doses
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 459 | 950 | 405 | 262
Doses | 5 [2.5 to 5] | 20 [15 to 20] | 10 [5 to 10] | 220 [220 to 300]

26. Primary Outcome: Number of Participants With Dose Reduction by Each OAC Treatment
Description: Baseline was defined as the time of index date which was defined as the first prescription with any of the oral anticoagulants, that is, participants with NVAF for the first time starting a therapy with any of the NOACs between 01-Jan-2013 and 30-Jun-2018.
Time Frame: From baseline (index date) until switch of treatment, discontinuation, death, first stroke/systemic embolism, or major bleeding, or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 459 | 950 | 405 | 262
Participants | 0 | 375 | 173 | 159

27. Primary Outcome: Time to Dose Reduction by Each OAC Treatment
Description: as for outcome 1
Time Frame: From index date until date of dose reduction or until end of follow-up, anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 106 | 32 | 10 | 10
Days | 68.5 [26.8 to 202.8] | 479 [144.8 to 725.2] | 523 [308.8 to 789.8] | 324 [103.5 to 1002.2]

28. Primary Outcome: Number of Participants With Treatment Discontinuation
Description: Discontinuation was defined as the first day of a period of at least 30 consecutive days in which 0 days' supply for the index OAC was detected. The date of discontinuation was the end date of the last filled prescription before the treatment gap. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: From index date until date of discontinuation, or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 78 | 147

29. Primary Outcome: Time to Discontinuation
Description: Time to discontinuation was defined as the number of days from the date of index oral anticoagulant prescription to the date of discontinuation. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: as for outcome 28
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 78 | 147
Days | 332 [130 to 679] | 463 [222 to 856]

30. Primary Outcome: Number of Participants According to Reasons for Discontinuation
Description: as for outcome 28
Time Frame: as for outcome 2
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 78 | 147
Participants
  Adverse drug reaction - not bleeding | 4 | 4
  Adverse drug reaction - any bleeding | 2 | 3
  Bleeding risk | 5 | 12
  Change to rhythm control | 1 | 2
  INR out of goal | 2 | 0
  No identifiable cause | 32 | 73
  NVAF improvement | 13 | 17
  Another event (acute myocardial infarction, worsening of renal failure, worsening of NVAF) | 7 | 11
  Participant preference | 10 | 20
  Problems related with drug access | 2 | 5

31. Primary Outcome: Number of Participants According to INR Measurements During Follow-up (Warfarin Group Only)
Description: as for outcome 1
Time Frame: From 1 Month to maximum 6.5 years (Jan 2013 to Jul 2019)
Population: Analysis population included all eligible participants diagnosed with NVAF who initiated treatment with warfarin and NOACs between 01-January-2013 to 30-June-2018 or who were exposed to warfarin before 2013 and initiated treatment with NOACs within the established period. This outcome measure was planned to be analyzed for the warfarin group only.
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin
Number analyzed (Participants) | 459
Participants
  0 | 54
  1 | 56
  2 | 53
  3 | 44
  4 | 34
  5 | 21
  6 | 28
  7 | 18
  8 | 16
  9 | 21
  10 | 13
  11 | 12
  12 or more | 89

32. Primary Outcome: Number of Participants Who Switched to Another OAC Treatment
Description: A switch among anticoagulants was defined as a prescription filled for non-index anticoagulants within +/- 30 days after the date of discontinuation. Index date was defined as the first prescription with OAC (i.e., warfarin or NOAC) for NVAF between 01-January-2013 to 30-June-2018.
Time Frame: From index date until switch of treatment or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 459 | 1617
Participants | 194 | 151

33. Primary Outcome: Time to Switch to Another OAC Treatment
Description: as for outcome 32
Time Frame: as for outcome 32
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 194 | 151
Days | 2309.0 [2274.7 to 2343.3] | 1114.0 [948.1 to 1279.9]

34. Primary Outcome: Number of Participants According to Reasons for Switching OAC Treatment
Description: as for outcome 32
Time Frame: From index date until switch of treatment, or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | NOACs
Number analyzed (Participants) | 194 | 151
Participants
  Adverse drug reaction - not bleeding | 2 | 16
  Adverse drug reaction - any bleeding | 0 | 3
  Bleeding risk | 7 | 5
  Drug interaction | 1 | 0
  INR out of goal | 65 | 0
  No identifiable cause | 112 | 87
  Another event (acute myocardial infarction, worsening of renal failure, worsening of NVAF) | 6 | 28
  Participant preference | 1 | 5
  Problems related with drug access | 0 | 7

35. Primary Outcome: Number of Participants With Concomitant Therapies by OAC Prescription
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- NOACs - Rivaroxaban: Participants diagnosed with NVAF, who initiated treatment with rivaroxaban between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated rivaroxaban between 01-January-2013 and 30-June-2018 were also included.
- NOACs - Apixaban: Participants diagnosed with NVAF, who initiated treatment with apixaban between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated apixaban between 01-January-2013 and 30-June-2018 were also included.
- NOACs - Dabigatran: Participants diagnosed with NVAF, who initiated treatment with dabigatran between 01-January-2013 and 30-June-2018 were observed in this retrospective study. Participants who were exposed to warfarin before 2013 and initiated dabigatran between 01-January-2013 and 30-June-2018 were also included.
Arm/Group | Warfarin | NOACs - Rivaroxaban | NOACs - Apixaban | NOACs - Dabigatran
Number analyzed (Participants) | 459 | 950 | 405 | 262
Participants
  Beta (β)-blockers | 305 | 641 | 270 | 186
  Statins | 266 | 598 | 266 | 164
  Angiotensin II receptor blockers | 232 | 543 | 247 | 164
  Furosemide | 126 | 275 | 98 | 61
  Angiotensin converting enzyme inhibitor | 119 | 182 | 71 | 50
  Proton pump inhibitor | 116 | 242 | 105 | 63
  Calcium channel blockers | 112 | 260 | 129 | 89
  Levothyroxine | 96 | 224 | 81 | 52
  Thiazide diuretics | 85 | 159 | 82 | 59
  Bronchodilators | 76 | 144 | 45 | 33
  Potassium sparing diuretic | 75 | 155 | 55 | 24
  Antiarrhythmics | 75 | 206 | 65 | 55
  Oral antidiabetics | 72 | 159 | 72 | 42

36. Primary Outcome: Number of Participants Who Were Previously Exposed to Warfarin (NOACs Group Only)
Description: as for outcome 1
Time Frame: Up to 6 months prior to index date
Population: Analysis population included all eligible participants diagnosed with NVAF who initiated treatment with warfarin and NOACs between 01-January-2013 to 30-June-2018 or who were exposed to warfarin before 2013 and initiated treatment with NOACs within the established period. This outcome measure was planned to be analyzed for the NOACs group only.
Measure: Count of Participants; unit: Participants
Arm/Group | NOACs
Number analyzed (Participants) | 1617
Participants | 181

ADVERSE EVENTS:
Time Frame: From index date until switch of treatment, discontinuation, death, first stroke/systemic embolism, or major bleeding, or until end of follow-up, whichever occurred first anytime between Jan 2013 to Jul 2019(approximately 6.5 years); retrieved data was analyzed during approximately 2 months of this observational study
Description: The study was a retrospective study of existing medical records and claim database; hence, only adverse events related to major bleeding were collected and reported. There was no specific medical dictionary utilized to record adverse events. Non-SAEs were not collected and reported.
Arm/Group | Warfarin | NOACs
All-Cause Mortality (participants affected / at risk) | 1/459 | 5/1617
Serious Adverse Events (participants affected / at risk) | 41/459 | 44/1617
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=459) | NOACs (N=1617)
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 19 | 23
Other major bleeding (Blood and lymphatic system disorders) | 17 | 19
Hemorrhagic cerebrovascular event (Blood and lymphatic system disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT04234698/Prot_SAP_000.pdf